CLINICAL TRIAL: NCT05945589
Title: Effects of Participatory Art-Based Activity On Health of Older Community-Dwellers: The Singapore Art-Health Randomized Control Trial Study
Brief Title: The Singapore Art-Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Collaborators: National Gallery Singapore, Singapore (Unknown); Sheffield Hallam University (Other); Université de Montréal (Other)
Responsible Party: Principal Investigator, Andy Hau Yan Ho, PhD, EdD, Principal Investigator, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-2020-02-005
Record Dates: First submitted 2023-07-05; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Art; Wellness, Psychological; Frailty; Quality of Life
Keywords: Art; Museum; Quality of Life; Frailty
MeSH Terms: conditions — Psychological Well-Being; Frailty

STUDY DESIGN:
Intervention Model Description: Intervention group participants will be invited to engaged in a 12-week participatory art program at the gallery. Participants in the control condition will not offered any art-based activities. All participants were advised not to participate in concurrent health art-based interventions during the research period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Simple randomization was administered by a dedicated research team member using an automated randomizer. Consenting participants were randomly assigned a number, where 1 = Intervention group, and 2 = Control group. Participants and other members of the research team were blinded to the randomization outcomes, and the outcome of the allocation was revealed after completion of the baseline assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Singapore A-Health Group (Experimental): A 12-week professionally led participatory art program at the gallery with each week comprising one 2-hour art session, totaling 24 hours of museum tours and participatory art activities.
  Interventions: Behavioral: Singapore A-Health Intervention
- Control Group (No Intervention): No art-based activities offered and advised not to participate in concurrent health and art-based interventions during the 12-week research period.

INTERVENTIONS:
Behavioral: Singapore A-Health Intervention — The Singapore A-Health Intervention spanned 12 weeks, with each weekly session lasting for two hours. The program is structured around three thematic domains of the past, present, and future. In each thematic domain consisting of four weeks, participants were tasked with creating an artwork related to the theme and incorporating the learned art techniques. The structure of each thematic domain follows the same structure: the first week involved a 45-minute docent-led gallery tour on three selected pieces of artworks, followed by a 75-minute artist-led brainstorming session where participants were introduced to the techniques and discuss ideas on the artwork to be created. The subsequent three sessions involved further guidance from the artist and a scaffolded delivery of art techniques for participants to incorporate their learning to their artwork. At the end of each domain, there was a showcase where participants present their artwork.
  Arms: Singapore A-Health Group

SUMMARY:
The goal of the Singapore Art-Health RCT is to examine the effect of a standardized 12-week museum -based participatory art program on health condition, well-being, and quality of life in older community dweller, one that adheres to the Montreal Art-Health framework with culturally specific modifications that are fitting to the local Singaporean context.

Participants will be randomized into an intervention group of a passive control group. Participants in the intervention group will be invited to participate in the 12-week Singapore Art-Health Intervention held at the National Gallery Singapore. All participants will be invited to complete four online psychometric assessments. Participants in the intervention group will be invited to completed an additional post-intervention survey and a feasibility focus group.

DETAILED DESCRIPTION:
Background: Population aging continues to be global health challenge. The prevalence of longstanding age-related conditions such as worsening physical, social, and mental health is expected to increase exponentially with a rapidly ageing population. The practice of participatory art in various settings has been found to be effective in the promotion, prevention and management of health and wellbeing conditions across the life span. However, its effect on health condition among the older population, particularly in the Asian context remains to be investigated. In Montreal, findings from a pilot study provided strong evidence to show that a 12-week, standardized "Art-Health" participatory art program had multidimensional positive effects on the health outcomes of older community dwelling participants including improvements in wellbeing, quality of life, and frail condition.

Current Proposal: The current research will adopt and modify the Montreal Art-Health participatory art framework with local cultural specificity (i.e. The Singapore Art-Health Intervention), and tests its effectiveness in healthy and wellness promotion among a sample of Singaporean older adults via a randomized control trial.

Research Design: The study adopts a participatory action research paradigm and a single-site, open-label Randomized Control Trial (RCT) design to develop and examine the effect of a standardized 12-week museum-based participatory art activity on health condition, wellbeing, and quality of life in older community dwellers.

Sampling and Randomization: Allowing for an attrition rate of 5% at follow-up, a target sample of 110 provides 90% power to detect an effect size of 0.55 (based on the results of the pilot study) between the intervention group and the control group at 5% level of significance (two-tailed test). Participants will be randomized into an intervention group of a passive control group. Participants in the intervention group will be invited to participate in the 12-week Singapore A-Health Intervention held at the National Gallery Singapore.

Intervention Design: The Singapore Art-Health Intervention will span 12 weeks, with each weekly session lasting for two hours. The program is designed to impart basic art appreciation skill (formal analysis in art) and art making techniques to participants through engagement with the collection at the museum.

Outcome measures and Data Analysis: All participants will be invited to complete four online psychometric assessments. Participants in the intervention group will be invited to completed an additional post-intervention survey and a feasibility focus group. For the quantitative data, between and within comparisons of outcomes will be conducted by mixed model analysis of variance (ANOVA), repeated measures ANOVA, and pairwise t-tests with Bonferroni correction. The focus group discussions will be analyzed using thematic analysis with a grounded theory approach to provide insights to the participant's experience and impact of the Singapore Art-Health Intervention.

Importance of Research: The current research will develop and test the effectiveness of a culturally-specific Art-Health participatory art program on health and wellness promotion among a sample of Singaporean older adults. Working collaboratively with the National Gallery Singapore in program development and implementation will serve to ensure program sustainability upon research completion. This collaboration will also foster practice and knowledge transfer to accelerate creative ageing in the local society. Moreover, the findings will contribute to an international RCT for evaluating a standardized participatory art framework to address the impact of population ageing. It will be a potential breakthrough in the development of an efficient art and museum program for older adults locally and internationally.

ELIGIBILITY:
Inclusion Criteria:

* individuals above the age of 60,
* fluent in English
* able to access the internet to complete the online psychometric assessments

Exclusion Criteria:

* unable to provide informed consent
* diagnosed with mental health conditions

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life (EQ5D) | Baseline
  Quality of life will be assessed by EuroQol-5D (EQ5D) which comprised of two parts: (1) 5-item scale on mobility, self-care, daily activities, pain, and depressive symptoms, (2) a visual analog scale of the participant's perceived health ranging from 0 (worst health) to 100 (best health one can imagine)
Change in Quality of Life (EQ5D) | 5-week follow-up
  Quality of life will be assessed by EuroQol-5D (EQ5D) which comprised of two parts: (1) 5-item scale on mobility, self-care, daily activities, pain, and depressive symptoms, (2) a visual analog scale of the participant's perceived health ranging from 0 (worst health) to 100 (best health one can imagine)
Change in Quality of Life (EQ5D) | 9-week follow-up
  Quality of life will be assessed by EuroQol-5D (EQ5D) which comprised of two parts: (1) 5-item scale on mobility, self-care, daily activities, pain, and depressive symptoms, (2) a visual analog scale of the participant's perceived health ranging from 0 (worst health) to 100 (best health one can imagine)
Change in Quality of Life (EQ5D) | 12-week follow-up
  Quality of life will be assessed by EuroQol-5D (EQ5D) which comprised of two parts: (1) 5-item scale on mobility, self-care, daily activities, pain, and depressive symptoms, (2) a visual analog scale of the participant's perceived health ranging from 0 (worst health) to 100 (best health one can imagine)
Mental Wellbeing (WEMWBS) | Baseline
  Mental Wellbeing will be assessed by Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS), a 14-item scale assessing various domains of wellbeing.
Change in Mental Wellbeing (WEMWBS) | 5-week follow-up
  Mental Wellbeing will be assessed by Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS), a 14-item scale assessing various domains of wellbeing.
Change in Mental Wellbeing (WEMWBS) | 9-week follow-up
  Mental Wellbeing will be assessed by Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS), a 14-item scale assessing various domains of wellbeing.
Change in Mental Wellbeing (WEMWBS) | 12-week follow-up
  Mental Wellbeing will be assessed by Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS), a 14-item scale assessing various domains of wellbeing.
Frailty (CESAM) | Baseline
  Frailty will be assessed by the Centre of Excellence on Longevity Self-administered Questionnaire (CESAM). It is a 20-item scale assessing multiple aspects of health such as drug intake, memory complaints, health service utilization, and activities of daily living.
Change in Frailty (CESAM) | 5-week follow-up
  Frailty will be assessed by the Centre of Excellence on Longevity Self-administered Questionnaire (CESAM). It is a 20-item scale assessing multiple aspects of health such as drug intake, memory complaints, health service utilization, and activities of daily living.
Change in Frailty (CESAM) | 9-week follow-up
  Frailty will be assessed by the Centre of Excellence on Longevity Self-administered Questionnaire (CESAM). It is a 20-item scale assessing multiple aspects of health such as drug intake, memory complaints, health service utilization, and activities of daily living.
Change in Frailty (CESAM) | 12-week follow-up
  Frailty will be assessed by the Centre of Excellence on Longevity Self-administered Questionnaire (CESAM). It is a 20-item scale assessing multiple aspects of health such as drug intake, memory complaints, health service utilization, and activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Andy HY Ho, PhD, EdD, Principal Investigator — Nanyang Technological University
Locations (1):
- Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
There are currently no plans o make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Beauchet O, Cooper-Brown LA, Hayashi Y, Deveault M, Ho AHY, Launay CP. Health benefits of "Thursdays at the Montreal Museum of Fine Arts": Results of a randomized clinical trial. Maturitas. 2021 Nov;153:26-32. doi: 10.1016/j.maturitas.2021.07.013. Epub 2021 Jul 31. PMID 34654525
- [Background] Beauchet O, Bastien T, Mittelman M, Hayashi Y, Hau Yan Ho A. Participatory art-based activity, community-dwelling older adults and changes in health condition: Results from a pre-post intervention, single-arm, prospective and longitudinal study. Maturitas. 2020 Apr;134:8-14. doi: 10.1016/j.maturitas.2020.01.006. Epub 2020 Jan 13. PMID 32143777
- [Derived] Ho AHY, Ma SHX, Tan MKB, Bajpai R, Goh SSN, Yeo G, Teng A, Yang Y, Galery K, Beauchet O. Effects of participatory 'A'rt-Based Activity On 'Health' of Older Community-Dwellers: results from a randomized control trial of the Singapore A-Health Intervention. Front Med (Lausanne). 2023 Dec 21;10:1238562. doi: 10.3389/fmed.2023.1238562. eCollection 2023. PMID 38188333